CLINICAL TRIAL: NCT00092027
Title: A Randomized, Double-Blind, Multicenter, Placebo-Controlled Study to Compare the Safety and Tolerability of an Oral Buffered Solution of Alendronate Sodium 70 mg Once-Weekly Versus Placebo for the Treatment of Osteoporosis in Postmenopausal Women
Brief Title: A Study to Evaluate the Safety and Tolerability of MK0217 in Women (0217-219)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0217-219; MK0217-219; 2004_017
Record Dates: First submitted 2004-09-21; First posted 2004-09-24 (Estimated); Last update posted 2024-08-14 (Actual); Status verified 2022-02

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Alendronate; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0217, alendronate sodium/Duration of Treatment: 6 months
Drug: Comparator: placebo / Duration of Treatment: 6 months

SUMMARY:
This study is to assess the safety and tolerability of MK0217 being evaluated to treat women with postmenopausal osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Women with postmenopausal osteoporosis

Exclusion Criteria:

* High risk for fractures
* Esophageal abnormalities
* Upper gastrointestinal symptoms that are not relieved with medication
* Metabolic bone disease (example - vitamin D deficiency)
* Medications that would affect the breakdown or build-up of bone

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2003-03-19 (Actual); Primary Completion 2004-03-15 (Actual); Study Completion 2004-03-15 (Actual)

PRIMARY OUTCOMES:
To evaluate the upper gastrointestinal (UGI) safety and tolerability of 6 months of treatment with once weekly alendronate 70 mg in an oral buffered solution in comparison to placebo in postmenopausal women with osteoporosis

SECONDARY OUTCOMES:
To evaluate the overall safety and tolerability of once weekly alendronate 70 mg oral buffered solution versus placebo
To evaluate the mean percent change from baseline in bone markers (BSAP, Urinary NTx) at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Cryer B, Binkley N, Simonelli C, Lewiecki EM, Lanza F, Chen E, Petruschke RA, Mullen C, de Papp AE. A randomized, placebo-controlled, 6-month study of once-weekly alendronate oral solution for postmenopausal osteoporosis. Am J Geriatr Pharmacother. 2005 Sep;3(3):127-36. doi: 10.1016/s1543-5946(05)80019-4. PMID 16257815